CLINICAL TRIAL: NCT06298565
Title: A Non-interventional, Post-authorisation Safety Study of Patients Treated With Efgartigimod Alfa
Status: Recruiting | Type: Observational
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Other Study IDs: ARGX-113-PASS-2208
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — efgartigimod alfa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- efgartigimod cohort: patients treated with efgartigimod
  Interventions: Biological: efgartigimod
- non-efgartigimod cohort: patient treated with other MG medication

INTERVENTIONS:
Biological: efgartigimod — efgartigimod
  Groups: efgartigimod cohort

SUMMARY:
This is a non-interventional, prospective, post authorization safety study. Patients with gMG who are expected to start treatment with efgartigimod at enrolment or are within their first cycle of efgartigimod at enrolment will be eligible to enroll into the efgartigimod cohort. Patients with gMG who have not been exposed to efgartigimod and for whom it is not planned to start treatment with efgartigimod at enrolment will be eligible to enroll into the non-efgartigimod cohort.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with gMG who are expected to start commercial efgartigimod at enrolment or who are within their first cycle of efgartigimod at enrolment or Patients diagnosed with gMG who have not been exposed to efgartigimod and for whom it is not planned to start treatment with efgartigimod at enrolment
* Have provided appropriate written informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with gMG
Sampling Method: Non-Probability Sample
Enrollment: 680 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2034-06 (Estimated); Study Completion 2034-06 (Estimated)

PRIMARY OUTCOMES:
The overall long-term safety of efgartigimod including the occurrence of serious infections in generalized myasthenia gravis (gMG) patients treated with efgartigimod compared to gMG patients not exposed to efgartigimod | up to 10 years

CONTACTS AND LOCATIONS:
Locations (35):
- United States (17):
  - UCSF Medical Center - Helen Diller Family Comprehensive Cancer Center - Brain Tumor Center,, San Francisco, California
  - SFM Clinical Research, LLC, Boca Raton, Florida
  - University of Florida College of Medicine Jacksonville, Jacksonville Beach, Florida
  - Medsol Clinical Research Center Inc, Port Charlotte, Florida
  - BayCare Health System, Inc. St Anthony's Hospital, St. Petersburg, Florida
  - Prairie Education and Research Cooperative and HSHS Medical Group, O'Fallon, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Norton Neuroscience Institute, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Oregon Health and Science University, Portland, Oregon
  - University of Colorado Hospital, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - National Neuromuscular Research Institute, Austin, Texas
  - BCN Research, LLC - Gamma Therapeutic Center, Greenfield, Wisconsin
- Kepler Universitätsklinikum, Universitätsklinik für Neurologie, Med Campus III, Linz, Austria
- UZ Leuven (University Hospitals Leuven), Leuven, Belgium
- Germany (7):
  - Klinikum Altenburger Land GmbH, Altenburg
  - St. Josef-Hospital Klinikum der Ruhr Universitaet Bochum, Bochum
  - Klinikum Christophsbad, Göppingen
  - Georg-August-Universität Göttingen, Göttingen
  - Klinikum Oberberg, Gummersbach
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Würzburg, Würzburg
- Italy (5):
  - Piazza OMS - Organizzazione Mondiale della Sanità, Bergamo
  - Ospedale Bellaria - Clinica Neurologica, Bologna
  - Azienda Ospedaliera di Rilievo Nazionale Cardarelli, Napoli
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
- Spain (4):
  - Hospital Universitari Vall d'Hebron, Unitat de Malalties Neuromusculars, Servei de Neurologia, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Clinico Universitario San Carlos, Madrid
  - Hospital Universitario Virgen Macarena, Seville

IPD SHARING:
Plan to Share IPD: Undecided